CLINICAL TRIAL: NCT05544162
Title: Personalized Targeted Nutrition Via StructurEd Nutrition Delivery Pathway to Improve Resilience in Older Adult Trauma Patients
Brief Title: Personalized Nutrition Delivery to Improve Resilience in Older Adult Trauma Patients
Acronym: SeND Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00110867
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Trauma; Critical Illness
MeSH Terms: conditions — Wounds and Injuries; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeND Home precision nutrition pathway (Experimental): Oral nutrition supplements (ONS) will be given, at maximum, three times per day throughout hospitalization. Upon discharge, participants will be given 4-weeks' worth of oral supplements to take. Adjustments may be made based on indirect calorimetry (IC) measurements by the clinical dietitian.
  Interventions: Dietary Supplement: Nutrition supplement - Ensure shakes
- Control pathway (No Intervention): Standard of care nutrition delivery throughout hospitalization. Upon discharge they will be sent home with standard nutrition information without Indirect Calorimetry (IC) guidance.

INTERVENTIONS:
Dietary Supplement: Nutrition supplement - Ensure shakes — Ensure shakes will be take up to 3 times a day throughout hospitalization and for 4 weeks after discharge.
  Arms: SeND Home precision nutrition pathway

SUMMARY:
This is a Pilot study designed to set up for an randomized clinical trial (RCT) comparing the SeND Home pathway to a standard of care nutrition delivery in critically ill older adult trauma patients. Subjects will be randomized 3:1 to either SeND Home precision nutrition pathway or control arm. Subjects randomized to the SeND Home arm will receive oral nutrition supplements (ONS) up to 3 times per day while in the hospital and for 4 weeks after discharge. Subjects in the standard of care arm will receive normal nutrition recommendations from their clinical providers. Participants in both groups will undergo non-invasive tests that measure how much energy (calories) they are using, body composition, and muscle mass.

DETAILED DESCRIPTION:
This is a Pilot study designed to set up for an randomized clinical trial (RCT) comparing the SeND Home pathway to a standard of care nutrition delivery in critically ill older adult trauma patients. The SeND Home Pathway supports patients from ICU admission to 2-weeks post-hospital discharge, providing a comprehensive and personalized plan of care carried to completion.

Subjects will be randomized 3:1 to either SeND Home precision nutrition pathway or control arm. Subjects randomized to the SeND Home arm will receive oral nutrition supplements (Ensure shakes) up to 3 times per day while in the hospital and for 4 weeks after discharge. Some subjects in this arm will be asked to participate in an interview after being discharged from the hospital. Subjects in the standard of care arm will receive normal nutrition recommendations from their clinical providers.

Participants in both groups will undergo non-invasive tests that measure how much energy (calories) they are using, body composition, and muscle mass. They will also be asked to complete walking and strength tests, and surveys about quality of life.These will be done every 3-7 days during hospitalization, at hospital discharge, and at a 3 month post-discharge follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 60 years old and admitted to the trauma service
* Patients who have had a standard of care CT scan

Exclusion Criteria:

* Expected withdrawal of life-sustaining treatment within 48 hours
* Prisoners
* Unable to provide informed consent
* Non-English speakers
* Traumatic Brain Injury
* Allergic to milk or soy ingredients (Common allergen in Ensure shakes).
* Pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of SeND Home pathway | 18 months
  Enrollment goal of 90%

SECONDARY OUTCOMES:
Acceptability of SeND Home pathway | 24 months
  Measured by interviewing enrolled subjects and stakeholders
Fidelity of SeND Home pathway | 18 months
  Measured by the proportion of interventions delivered per protocol with a goal of 80%

CONTACTS AND LOCATIONS:
Overall Officials: Krista Haines, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT05544162/ICF_000.pdf